CLINICAL TRIAL: NCT00488332
Title: An Exploratory Study on Optical Assessment of Oral Mucositis
Status: Terminated | Type: Observational
Why Stopped: Terminated due to slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2005-0872
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Head and Neck Cancer; Oral Mucositis
Keywords: Head and Neck Cancer; Oral Mucositis; Optical Coherence Tomography; Fluorescence Spectroscopy; Optical Assessment
MeSH Terms: conditions — Head and Neck Neoplasms; Stomatitis | interventions — Tomography, Optical Coherence; Spectrometry, Fluorescence; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OCT + FS + Questionnaire: Optical Coherence Tomography (OCT) + Fluorescence Spectroscopy (FS) and Questionnaire
  Interventions: Procedure: Optical Coherence Tomography; Procedure: Fluorescence Spectroscopy; Behavioral: Pain Scale Questionnaire

INTERVENTIONS:
Procedure: Optical Coherence Tomography — Before radiation treatment and once a week thereafter.
  Other Names: OCT
Procedure: Fluorescence Spectroscopy — Before radiation treatment and once a week thereafter.
  Other Names: FS
Behavioral: Pain Scale Questionnaire — Administered before the examination, OCT, and FS and immediately afterward.
  Other Names: Survey

SUMMARY:
Objectives:

1. To assess the tolerability of performing optical coherence tomography and/or optical spectroscopy in patients with acute oral mucositis.
2. To determine the feasibility of obtaining optical coherence tomography images and/or fluorescence excitation emission matrices from normal and affected sites in patients with acute oral mucositis.
3. To compare optical data obtained with optical coherence tomography and/or spectroscopy with the clinical appearance and scoring of oral mucositis lesions.

DETAILED DESCRIPTION:
Optical coherence tomography (OCT) works similarly to ultrasound but uses infrared light waves rather than sound waves to create high-resolution pictures. This tool has been approved by the Food & Drug Administration (FDA), is used routinely for standard diagnosis of eye conditions, and is now being used to look inside your mouth for tissue changes.

For the OCT procedure, a small probe, about the size of a pencil eraser, will be gently placed against the lining of your mouth and light will be shone through the probe to create pictures of the tissue. The probe will be placed on 1-2 abnormal-looking areas and 1 normal-looking area inside the mouth. If there are no abnormal-looking areas, researchers will place the probe and make pictures of an area on the inside of the cheek and side of the tongue, since these are the areas most often affected by the chemotherapy and radiation therapies.

In fluorescence spectroscopy (FS), a small beam of light, shines through a small probe onto the lining of the mouth. A small amount of light will be emitted from the tissue in the form of fluorescence, similar to "glow in the dark" toys . This light is not seen by the eye, but it is detected by the probe and recorded by a computer.

For the FS procedure, a small probe, about the size of a pencil eraser, will be gently placed against the lining of your mouth and light will be shone through the probe. The probe will then collect the fluorescence light signals and they will be recorded on a computer. The probe will be placed on 1-2 abnormal-looking areas and 1 normal-looking area inside the mouth. If there are no abnormal-looking areas, researchers will place the probe and make pictures of an area on the inside of the cheek and side of the tongue, since these are the areas most often affected by the chemotherapy and radiation therapies.

If you agree to take part in this study, your mouth will be examined before your treatment begins, and then once a week after that. Every week, you will also be asked how much pain you are having on a scale of 1-10.

Photographs will be taken of the inside of the mouth with a standard camera. You will not be identified in these photographs.

You will be asked to return once a week until you finish all radiation treatments to have all the exams repeated. Most radiation treatments last about 6-8 weeks.

This is an investigational study. About 18 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients greater than 18 years old.
2. Patients undergoing radiation therapy or chemoradiotherapy for head and neck cancer treatment.
3. Subject must sign an informed consent indicating awareness of the investigational nature of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals, minimally 18 years old, undergoing radiation therapy or chemoradiotherapy for head and neck cancer treatment.
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2006-03; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Optical assessment of oral mucositis in patients undergoing radiation or chemoradiation for head and neck cancer treatment | Two sets of oral scans; one at baseline and the second 2 weeks into therapy

CONTACTS AND LOCATIONS:
Overall Officials: Ann M. Gillenwater, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org